CLINICAL TRIAL: NCT05466552
Title: A Prospective Multinational Registry on Preventive Left Ventricular Support With Impella in Anatomically High-risk PCI Treated Patients
Brief Title: The PROTECT-EU Study
Status: Recruiting | Type: Observational
Sponsor: Fondazione GISE Onlus (Other)
Collaborators: Abiomed Inc. (Industry); University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: GISE_PROTECTEU
Record Dates: First submitted 2022-05-25; First posted 2022-07-20 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: High-risk PCI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PCI procedure — During the PCI procedure, use of ECMO/Impella 5.0 is allowed hemodynamic instability (bail- out).

SUMMARY:
The PROTECT-EU Registry is a prospective, non-randomized, multi-national registry to evaluate 90 days outcomes in high risk-PCI (Percutaneous coronary intervention) patients treated with a preventive strategy with Impella CP® System.

DETAILED DESCRIPTION:
The PROTECT-EU Registry is a prospective multinational registry on preventive left ventricular support with Impella in high-risk PCI treated patients. The aim is to confirm and improve the Impella effectiveness in a selected all comers high risk population undergoing supported HR-PCI (high risk-PCI) with Impella implantation before PCI.

ELIGIBILITY:
Inclusion Criteria:

Patients with non-emergent chronic or acute coronary syndromes (the former refused from surgical revascularization) with reduced LVEF (left ventricular ejection fraction)(<=40%) and indication for high-risk PCI AND

Intended high-risk PCI defined as having at least one of the following criteria:

* Unprotected left main distal disease involving bifurcation or trifurcation or left main equivalent
* Diffuse degenerated (>5 mm) saphenous vein grafts involving the proximal or distal anastomosis or in-stent restenosis
* LAD (left anterior descending) long lesions (>48 mm) involving both septal and diagonal branches requiring multiple and overlapping stents
* Diffuse and severely calcified lesions (see protocol definition) with need for debulking devices (directional, rotational, orbital, and laser)
* Last patent conduit
* Complex CTO (chronic total occlusion) (J-CTO score 3) or CTO in patients with MVD (Coronary Microvascular Disease)
* MV-PCI (Multivessel Percutaneous Coronary Intervention) in patient with a Syntax score>32 undergoing planned complete revascularization (see protocol definition of severe stenosis)
* (only in ACS Acute Coronary Syndrome patients) Giant thrombus (length ≥3x vessel diameter) in the context of MVD or Syntax score >32.

Exclusion Criteria:

* Classic CS Coronary Sinus (relative hypotension as SBP < 90 mmHg, or MAP <60 mmHg or >30 mmHg drop from baseline and drugs/device used to maintain blood pressure above these targets and/or symptoms/signs of hypoperfusion as cardiac index <2.2, lactate ≥ 2mmol/L (24).
* Cardiac arrest
* Patients admitted for ACS due to ST-elevation MI (ST Elevation Myocardial Infarction)
* Contraindication to Impella positioning: mural thrombus in the left ventricle; presence of a mechanical aortic valve; severe aortic stenosis or valvular regurgitation; severe peripheral arterial disease precluding placement of the Impella System; haematological disorder causing fragility of the blood cells or hemolysis; hypertrophic obstructive cardiomyopathy (HOCM); aneurysm or severe anomaly of the ascending aorta and/or aortic arch; significant right heart failure; presence of an atrial or ventricular sepal defect (including post-infarct VSD Ventricular Septal Defect); left ventricular rupture; cardiac tamponade; recent TIA or stroke (within 1 month); contraindication to anticoagulation
* Age < 18 or > 80 years old
* Inability to understand and sign informed consent
* Serious known concomitant disease with a life expectancy of less than one year
* Prior thrombolytic therapy during the index event (within 72 h of presentation)
* Severe renal impairment Renal insufficiency (GFR Glomerular Filtration Rate <30 ml/min)
* Patients on oral anticoagulation therapy (including novel oral anticoagulant such as dabigatran, rivaroxaban, apixaban and edoxaban) at the time of PCI
* Suspected or known pregnancy
* Suspected active infection
* Current participation in an investigational study using a drug or device.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: High-risk PCI population defined with clinical and angiographic criteria. Impella will be started after coronary angiography and before PCI and will be discontinued before discharge from the catheterization laboratory if the patient is deemed hemodynamically stable. All subjects will have 1-year follow-up. The primary endpoint will be assessed at 90 days follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 859 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Death | at 90 days
  Composite endpoint of all-cause death
Cerebrovascular accident | at 90 days
  Cerebrovascular accident at 90 days
infarction | at 90 days
  myocardial infarction
revascularization | at 90 days
  repeat revascularization

SECONDARY OUTCOMES:
hospitalization for cardiovascular cause | at 90 days
  cardiovascular disease
hospitalization for cardiovascular cause | at 1 year
  cardiovascular disease
cerebrovascular events | at 90 days
  cerebrovascular events (all, stroke and TIA)
cerebrovascular events | at 1 year
  cerebrovascular events (all, stroke and TIA)
QoL: KCCQ | at 90 days
  KCCQ (Kansas City Cardiomyopathy Questionnaire)
QoL: EQ-5D | at 90 days
  EQ-5D: EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys.
QoL: KCCQ | at 1 year
  KCCQ (Kansas City Cardiomyopathy Questionnaire)
QoL: EQ-5D | at 1 year
  EQ-5D: EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No